CLINICAL TRIAL: NCT04752306
Title: The Integration of Sensor Technology in Disposable Pads: a Needs Assessment in Nursing Homes
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: BC-07270
Record Dates: First submitted 2020-10-13; First posted 2021-02-12 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2020-10

CONDITIONS: Incontinence
Keywords: incontinence; pads; sensor technology
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- residents: 10 residents
  * Minimum 1x > 1week had experience with incontinence material
  * MMSE score >23
  * good verbal communication
  Interventions: Other: Interviews
- healthcare workers: 8 healthcare workers working in setting, no exclusion criteria
  Interventions: Other: Interviews
- policymakers: 2 policymakers responsible for the purchase of incontinence material
  Interventions: Other: Interviews

INTERVENTIONS:
Other: Interviews — Semi-structured interviews will take place between June and August 2020. Eight individual interviews with healthcare workers, ten individual interviews with residents and two individual interviews with policymakers. Interviews with the healthcare workers and policymakers will take place in a meeting room at the nursing home of employment. One interview with a policymaker will take place online. Interviews with residents will be hold in their personal room.

SUMMARY:
The aim of the study is to explore the criteria and conditions for the integration of sensor technology in disposable pads according to the needs and opinions of residents with incontinence, healthcare workers, and policymakers in nursing homes.

ELIGIBILITY:
Inclusion Criteria:

* Residents

  1. if they have worn absorbent incontinence products minimum one time for more than one week
  2. if they have a Mini-Mental State Examination (MMSE)-score of >23
  3. if they are able to communicate verbally
* Health care workers
* if they are health care assistants or nurses
* Policymakers if they have a role in the financial decisions regarding incontinence material.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 10 residents, 8 healthcare workers and 2 policymakers from 3 nursinghomes in Flandres (Belgium)
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
requirements for sensor technology in disposable bodyworns measured with a semi-structured questionnaire | 6 months
  To successfully implement sensor technology; requirements for the sensor technology must be defined according to the relevant stakeholder groups. Throughout the development process the researcher will question nursing home residents, healthcare workers and policymakers in semi-structured interviews to identify how the sensor technology could improve the quality of care, and reduce workload and costs.

CONTACTS AND LOCATIONS:
Locations (3):
- Belgium (3):
  - Residentie Vroonstalle, Ghent, Oost-vlaanderen
  - Rustenhove, Ledegem, West-Vlaanderen
  - Residentie Brugse Vaart, Ghent

IPD SHARING:
Plan to Share IPD: Undecided
Data will be available upon request

REFERENCES:
- [Derived] Raepsaet C, Serraes B, Verhaeghe S, Beeckman D. Integrating Sensor Technology in Disposable Body-Worn Absorbent Products: A Qualitative Study to Define User Profile, (Technical) Criteria, Conditions, and Potential Benefits. J Wound Ostomy Continence Nurs. 2021 Nov-Dec 01;48(6):560-567. doi: 10.1097/WON.0000000000000812. PMID 34781313